CLINICAL TRIAL: NCT04298827
Title: Optimizing Prehabilitation in Gynecologic Oncology
Brief Title: Gyn Onc Prehab Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Shannon Grabosch, MD, Assistant Professor of Gynecologic Oncology, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30334
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Gynecologic Cancer; Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Surgery; Treatment Adherence; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unimodal (Active Comparator): Patients will be randomized at their pre-surgical consultation. Patients will undergo a physical therapy evaluation prior to surgery and at 4 and 8 weeks post-op. Their preoperative visits will be as close to 4 weeks before surgery as possible but given the urgency of some of these surgeries and diagnoses, treatment will not be delayed to complete the components of this study. The patient will also be asked to complete a quality of life assessment at the beginning and end of the study as well as an anonymous survey at the conclusion of the study evaluating her satisfaction with the experiment.
  Interventions: Other: Unimodal
- Trimodal (Active Comparator): Patients will be randomized at their pre-surgical consultation. Patients will undergo a physical therapy evaluation, nutritional counseling and group therapy, prior to surgery and at 4 and 8 weeks post-op. Their preoperative visits will be as close to 4 weeks before surgery as possible but given the urgency of some of these surgeries and diagnoses, treatment will not be delayed to complete the components of this study. The patient will also be asked to complete a quality of life assessment at the beginning and end of the study as well as an anonymous survey at the conclusion of the study evaluating her satisfaction with the experiment. Patient nutritional assessments will be obtained with Patient Generated Subjective Global Assessment questionnaires as well as targeted questioning by the dietician.
  Interventions: Other: Trimodal

INTERVENTIONS:
Other: Unimodal — Patients will receive physical therapy alone.
  Arms: Unimodal
Other: Trimodal — Patients will receive physical therapy, nutrition counseling, and cognitive behavioral therapy in the form of group counseling.
  Arms: Trimodal

SUMMARY:
Patients will be randomized to a unimodal or trimodal prehabilitation program prior to surgery for known or suspected gynecologic cancer.

DETAILED DESCRIPTION:
Prehabilitation generally refers to the act of an intervention prior to a known potentially debilitating event. Usually taking the form of physical therapy prior to surgery, prehabilitation programs have demonstrated success in colorectal, urological, and surgical oncology cases. Patients with a gynecologic oncology diagnosis face an arduous course. Their treatment generally involves a major surgery and is often followed by chemotherapy, radiation, or both.The patient population is generally older in life as the average age for an endometrial or ovarian cancer diagnosis is 63. These patients may already have a lower performance status at baseline deeming their treatment course exponentially more difficult to endure. Women with gynecologic cancer suffer significant mental duress often living in fear of the high rates of recurrence from some of these malignancies suggesting they may benefit from psychologic support and counseling through their treatment.

Given the proven success in other surgical disciplines, we believe that instituting prehabilitation programs should be standard of care. Patients will be randomized to a trimodal approach (physical therapy, nutritional counseling, cognitive behavioral therapy) versus a unimodal intervention (physical therapy) for a formal prehabilitation program. Our primary outcome will be functional return to baseline following surgery with secondary outcomes including items such as quality of life assessments, patient satisfaction, and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patient who will be undergoing a planned surgery for known or presumed gynecologic cancer diagnosis.

Exclusion Criteria:

* Non-English speaking patients
* Surgeries done for palliative intent
* Poor performance status or other inability to participate in physical therapy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | During the approximate 12 week study period
  Patients will have a preoperative physical therapy assessment incorporating standard evaluations of a 6 minute walk test, grip strength, and timed up and go. These will serve as the individual patient's baseline for subsequent comparison after surgery.
Six Minute Walk Test | During the approximate 12 week study period
  Patients will have a preoperative physical therapy assessment incorporating standard evaluations of a 6 minute walk test, grip strength, and timed up and go. These will serve as the individual patient's baseline for subsequent comparison after surgery.
Grip Strength | During the approximate 12 week study period
  Patients will have a preoperative physical therapy assessment incorporating standard evaluations of a 6 minute walk test, grip strength, and timed up and go. These will serve as the individual patient's baseline for subsequent comparison after surgery.

SECONDARY OUTCOMES:
Readmission Rates | During the 8 weeks after surgery (12 week approximate total study period)
  Need for postoperative readmission with be monitored in each group.
Complication Rates | During the 12 week approximate total study period
  Surgical or treatment complications with be monitored in each group.
Patient Satisfaction | At the conclusion of the approximate 12 week study period
  Patients from each group will be asked to complete an anonymous survey evaluating their satisfaction with the program.
Quality of Life FACT-G Assessment | During the 12 week approximate total study period
  Patients will complete baseline and follow up quality of life assessments using the FACT-G (Functional Assessment of Cancer Therapy-General). This is a 28 question quality of life assessment with scores ranging from 0 to 112 (higher scores correlate with a higher quality of life).
Treatment Completion | At the conclusion of the 12 week approximate total study period
  Rate of program completion will be assessed for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Grabosch, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside of members of the research team.